CLINICAL TRIAL: NCT04434456
Title: Prospective Observational Study of CGuard MicroNet Covered Stent System Use as a Flow Diverter in the Endovascular Exclusion of Carotid Artery Aneurysms. (CGuard Divert-and-HEAL C-HEAL)
Brief Title: Carotid Artery Aneurysm Treatment Using CGuard Divert-And-Heal Strategy
Acronym: C-HEAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: John Paul II Hospital, Krakow (Other)
Responsible Party: Sponsor
Other Study IDs: C-HEAL
Record Dates: First submitted 2020-06-08; First posted 2020-06-16 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Carotid Artery Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CGuard stenting (interventional): CGuard implantation in the carotid artery with aneurysm requiring intervention
  Interventions: Device: CGuard stent implantation

INTERVENTIONS:
Device: CGuard stent implantation — CGuard stent implantation in the carotid artery with symptomatic, dissecting or enlarging aneurysm

SUMMARY:
Non-randomized, single arm, open label, academic observational study of CGuard MicroNet covered stent system use to achieve endovascular lumen reconstruction in carotid artery aneurysms with indications for treatment (enlarging and/or dissecting / symptomatic).

Jagiellonian University Medical College research project.

DETAILED DESCRIPTION:
Carotid artery aneurysm (CAA) is a relatively infrequent, but significant clinical condition with numerous diagnostic and therapeutic implications. CAA affects laminal flow in the carotid artery implicating the risk of thrombus formation in the aneurysm cavity, and subsequent ischemic stroke from distal embolization. Another important clinical problem related to the CAA is a possible aneurysm dissection and rupture. Symptomatic CAA and increasing dimensions of CAA institute unquestioned indications for the CAA treatment.

Surgical carotid aneurysm repair bears a significant risk (periprocedural stroke, cranial nerve damage, carotid artery ligation). Therefore endovascular techniques of CAA exclusion were developed. Covered stents, stent-grafts, and combined stenting and aneurysm embolization with coils were applied. However, covered stents were demonstrated to increase the restenosis risk, and other complications such as CAA neck endo-leak.

Newer technique involves the flow diversion by implantation of stent in dense-structured stent (such as Wallstent) or stent-in-stent implantation. In this case a luminary flow dominates over aneurysm filling, which is limited by stent structure. Gradual thrombosis and occlusion of aneurysm cavity and healing of aneurysm follows.This method disadvantage was related to necessity of double stent load and increased restenosis risk (double metal layer).

These issues were addressed only recently by the double layer mesh stents that demonstrate natural flow diverting capabilities. CGuard Stent system is a self-expandable stent covered with PET mesh (MicroNet) that prevents plaque protrusion into the vessel lumen. In addition, in low flow conditions MicroNet can act as the flow diverter. These stents are routinely implanted in elevated risk plaques in high reference centers in Europe.

Several published observations indicate the CGuard stent also demonstrates flow-diverting capabilities, but the systematic observation of such application was not performed.

C-HEAL is a non-randomized, single arm, open label academic observational study of CGuard stent implantation in carotid arteries in patients with symptomatic, dissecting or enlarging carotid artery aneurysm. Procedures are performed according to the center routine, with application of proximal or distal embolic protection device (if feasible), and standard pharmacotherapy according to the current guidelines.

ELIGIBILITY:
General

Inclusion Criteria:

* Patients older than 18 years, eligible for endovascular carotid artery aneurysm treatment with Micronet covered stent per Vascular Team evaluation, according to local standards
* Written, informed consent to participate
* Agreement to attend protocol required (standard) follow up visits and examinations

Exclusion Criteria:

* Preferred treatment other than stenting (surgery or conservative treatment / observation) per Vascular Team evaluation
* Life expectancy <1 year (e.g. active neoplastic disease).
* Chronic kidney disease with creatinine > 3.0 mg/dL.
* Myocardial infarction in 72 hours proceeding the stenting procedure (if possible, postponing the procedure)
* Pregnancy (positive pregnancy test)
* Coagulopathy.
* History of uncontrolled contrast media intolerance

Angiographic

Inclusion Criteria:

* Carotid artery aneurysm confirmed on angiography - symptomatic, dissected or enlarging
* Aneurysm eligible for endovascular treatment per Vascular Team evaluation (according to current standards, guidelines and study center practice)

Exclusion Criteria:

* Unsuccessful true lumen engagement
* Aneurysm neck anatomy precluding healthy-to-healthy coverage with stent
* Anatomic variants precluding stent implantation
* Mobile (free-floating) plaque elements in aorta or arteries proximal to target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 to 25 patients meeting inclusion and exclusion criteria and evaluated by Vascular Team to receive an endovascular treatment for carotid artery aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of successful aneurysm exclusion | 6 months
  Successful aneurysm cavity exclusion and endovascular lumen reconstruction on routine, non-invasive CT angiography

SECONDARY OUTCOMES:
Rate of procedural success | Peri-procedural
  Procedural success defined as: Technical success (successful MicroNet covered stent delivery and implantation with complete aneurysm necks coverage) and Clinical success (no complications)
Rate of In-hospital MACNE (major adverse cardiac and neurological events) | 48 hrs or until discharge
  In-hospital MACNE (death, stroke, myocardial infarction)
MACNE at 30 days | 30 days
  MACNE at 30 days (death, stroke, myocardial infarction)
Number of peri-procedural complications | 48 hrs or until discharge
  Any complications occurring up to 48 hours post procedure
Rate of clinical efficacy at 6 months | 6 months
  Clinical efficacy defined as successful aneurysm exclusion and no procedure related complications
Rate of clinical efficacy at 12 months | 12 months
  Clinical efficacy defined as successful aneurysm exclusion and no procedure related complications
Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) in the target vessel segment | 6 months
  Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) in ultrasound evaluation of target vessel segment (if amenable to duplex Doppler examination)
Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) in target vessel segment | 12 months
  Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) in ultrasound evaluation of target vessel segment (if amenable to duplex Doppler examination)
Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) in target vessel segment | 24 months
  Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) in ultrasound evaluation of target vessel segment (if amenable to duplex Doppler examination)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Musialek, MD, DPhil, Principal Investigator — The John Paul II Hospital
Locations (1):
- Department of Cardiac and Vascular Diseases, The John Paul II Hospital, Krakow, Maloplska, Poland

IPD SHARING:
Plan to Share IPD: No